CLINICAL TRIAL: NCT03514888
Title: A Pilot Study for Hyperthermic Intraperitoneal Chemotherapy After Radical Cystectomy With Pelvic Lymph Node Dissection for High Risk Invasive Bladder Cancer
Brief Title: HIPEC After Radical Cystectomy for High Risk Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1708018468
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Invasive Bladder Cancer
Keywords: High-risk bladder cancer; Urothelial cancer; HIPEC; Mitomycin
MeSH Terms: interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Intervention Model Description: HIPEC with Mitomycin-C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIPEC after Radical Cystectomy (Experimental): After completion of radical cystectomy, HIPEC will be administered using closed abdomen technique for a duration of 60 minutes.
  Interventions: Procedure: HIPEC

INTERVENTIONS:
Procedure: HIPEC — 40mg of Mitomycin-C dissolved in 100ml normal saline will be added into the perfusate and instilled into the patient for a total of 60 minutes. After 60 minutes, the abdomen will be irrigated with 3 liters of normal saline.
  Other Names: Hyperthermic intraperitoneal chemotherapy

SUMMARY:
This is a non-randomized, non-blinded, pilot study administering hyperthermic intraperitoneal chemotherapy with Mitomycin-C in 10 men and women with muscle-invasive urothelial carcinoma of the bladder undergoing radical cystectomy with pelvic lymph node dissection who have risk factors for tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Primary urothelial cell carcinoma of the bladder
2. Patient's aged 45-85, both genders.
3. ECOG performance status < 1
4. Hematology: ANC > 1.5x109/L; Platelets > 100x109/L
5. Women with child bearing potential who are negative for pregnancy test (urine or blood) and who agree to use effective contraceptive method. Reliable contraception should be used from trial screening and must be continued throughout the study. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant.
6. Signed and dated written informed consent to participate in this clinical trial must be obtained prior to any study procedure.

   Either any of the following preoperative factors for increased risk of recurrence:
7. Lymphovascular invasion
8. Variant histology in the background of primary urothelial (notably plasmacytoid)
9. Clinical T3 or greater
10. Clinical N+
11. No prior neoadjuvant chemotherapy (NAC) or lack of response to NAC

    Or any of the following perioperative factors for increased risk of recurrence:
12. Palpable concern for extravesical disease
13. Tumor spillage/bladder entry
14. Suspicious nodes or positive intraoperative frozen sections

Exclusion Criteria:

1. Subjects who have previously undergone intraperitoneal chemotherapy.
2. Subjects with tumor histology other than urothelial cell carcinoma.
3. Patients on concurrent anti-cancer therapy other than that allowed in the study.
4. Other prior malignancies, except for cured non-melanoma skin cancer or curatively treated in situ carcinoma of the cervix or adequately treated malignancies for which there has been no evidence of activity for more than 3 years.
5. Subjects with renal insufficiency defined as creatinine > 1.5x the upper limit of normal or a calculated creatinine clearance of < 50 cc/min.
6. Subjects with a condition which may interfere with the subjects' ability to understand the requirements of the study.
7. Known HIV, Hepatitis B or Hepatitis C positive.
8. Subjects with uncontrolled concurrent illness including, but not limited to, ongoing or severe infection requiring antibiotics, symptomatic congestive heart failure, unstable angina pectoris, acute gastrointestinal bleeding, psychiatric illness or other condition which in the opinion of the investigator, places the patient at an unacceptable risk for participation in the study.
9. Any condition that would preclude the ability to deliver appropriate IP therapy.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Treatment toxicity | 90 days
  Treatment toxicity will be analyzed using NCI Common Terminology Criteria for Adverse Events-Version 4.0. Descriptive statistics will be used to determine proportion of grade III/V treatment toxicity. Expected grade III/V toxicity in surgical patients without HIPEC would be 3 out of 10 patients. With the addition of HIPEC, there would be a significant difference (p=0.05) if 6 out of 10 patients experienced a grade III/V toxicity. Therefore, if less than 6 patients experience a grade III/V we would consider this a "negative" finding.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas S Scherr, MD, Principal Investigator — Weill Cornell Medicine - New York Presbyterian Hospital
Locations (1):
- Weill Cornell Medicine - New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No